CLINICAL TRIAL: NCT04125342
Title: Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation in Obese or High-Risk Patients. A Randomized Clinical Trial.
Brief Title: Postextubation High-flow Therapy vs Noninvasive Ventilation in Obese or at High-risk Patients
Acronym: HINFOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Virgen de la Salud (Other)
Responsible Party: Principal Investigator, Gonzalo Hernandez Martinez, Study Chair, Hospital Virgen de la Salud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25/9/2019 nº17
Record Dates: First submitted 2019-10-03; First posted 2019-10-14 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Extubation Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conditioned NIV in High Risk Patients (Experimental)
  Interventions: Device: Preventive Conditioned NIV Therapy after planned extubation
- HFOT in High Risk Patients (Active Comparator)
  Interventions: Device: Preventive HFOT after planned extubation
- Conditioned NIV in Obese Intermediate Risk Patients (Experimental)
  Interventions: Device: Preventive Conditioned NIV Therapy after planned extubation
- HFOT in Obese Intermediate Risk Patient (Active Comparator)
  Interventions: Device: Preventive HFOT after planned extubation

INTERVENTIONS:
Device: Preventive Conditioned NIV Therapy after planned extubation — Conditioned NIV during 48 hours following extubation.
  Arms: Conditioned NIV in High Risk Patients; Conditioned NIV in Obese Intermediate Risk Patients
Device: Preventive HFOT after planned extubation — HFOT set according to patients tolerance during 48 hours following extubation
  Arms: HFOT in High Risk Patients; HFOT in Obese Intermediate Risk Patient

SUMMARY:
The main aim is to demonstrate whether reintubation rate is lower with preventive conditioned noninvasive ventilation (NIV) rather than with High-flow oxygen therapy (HFOT) in obese intermediate-risk patients and in high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

1. High-Risk Patients: Patients under mechanical ventilation for more than 24 hours considered at high risk according to the presence of more than 3 of the following risk factors:

   * >65 years.
   * Cardiac failure as the primary indication of mechanical ventilation.
   * Moderate to severe chronic obstructive pulmonary disease.
   * APACHE II >12 points the extubation day.
   * Body mass index >30.
   * Inability to manage respiratory secretions.
   * Not simple weaning.
   * More than 1 comorbidity.
   * More than 7 days under mechanical ventilation.
   * Hypercapnia during the spontaneous breathing trial.
   * Airway patency problems.
2. Obese Intermediate Risk Patients: Patients under mechanical ventilation for more than 24 hours with a Body mass index >30 and considered at intermediate risk according to the presence of less than 3 of the following risk factors:

   * >65 years.
   * Cardiac failure as the primary indication of mechanical ventilation.
   * Moderate to severe chronic obstructive pulmonary disease.
   * APACHE II >12 points the extubation day.
   * Inability to manage respiratory secretions.
   * Not simple weaning.
   * More than 1 comorbidity.
   * More than 7 days under mechanical ventilation.
   * Airway patency problems.

Exclusion Criteria:

* <18 years.
* Thacheotomized patients.
* Contraindications for NIV (recent facial or cervical trauma/surgery, active gastro-intestinal bleeding, lack of cooperation).
* Unscheduled extubation.
* Do not reintubate orders.
* No informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Reintubation rate | 7 days

SECONDARY OUTCOMES:
Intensive Care Unit mortality rate | 3 months
Hospital mortality rate | 3 months
Intensive Care Unit length of stay | 3 months
Hospital length of stay | 6 months
Respiratory infection rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Hernandez, Study Chair — SESCAM
Locations (2):
- Spain (2):
  - Hospital Virgen de la Salud, Toledo, Castille-La Mancha
  - La princesa University Hospital, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hernandez G, Dianti J, Paredes I, Moran F, Marquez M, Calle A, Colinas L, Alonso G, Carneiro P, Morales G, Suarez-Sipmann F, Canabal A, Goligher E, Roca O. Humidified Noninvasive Ventilation versus High-Flow Therapy to Prevent Reintubation in Patients with Obesity: A Randomized Clinical Trial. Am J Respir Crit Care Med. 2025 Feb;211(2):222-229. doi: 10.1164/rccm.202403-0523OC. PMID 39514845
- [Derived] Hernandez G, Paredes I, Moran F, Buj M, Colinas L, Rodriguez ML, Velasco A, Rodriguez P, Perez-Pedrero MJ, Suarez-Sipmann F, Canabal A, Cuena R, Blanch L, Roca O. Effect of postextubation noninvasive ventilation with active humidification vs high-flow nasal cannula on reintubation in patients at very high risk for extubation failure: a randomized trial. Intensive Care Med. 2022 Dec;48(12):1751-1759. doi: 10.1007/s00134-022-06919-3. Epub 2022 Nov 18. PMID 36400984